CLINICAL TRIAL: NCT03407469
Title: Measurement of Adherence and Health-related Quality of Life, and Health-Care Resource Utilization During Anticoagulation Therapy in Cancer-Related Venous Thromboembolism (VTE)
Brief Title: Measurement of Adherence and Health-Related Quality of Life, and Health-Care Resource Utilization
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0303; NCI-2018-00900 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer-related Venous Thromboembolism
Keywords: Questionnaires; Surveys; Cancer-related Venous Thromboembolism; VTE
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires: Questionnaires completed at the time participant joins this study and then about 30 days, 3 months, 6 months, and 12 months after that. Questionnaires will be about quality of life and experiences with treatment for venous thromboembolism (VTE).
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed at the time participant joins this study and then about 30 days, 3 months, 6 months, and 12 months after that. Questionnaires will be about quality of life and experiences with treatment for venous thromboembolism (VTE). It should take less than 10 minutes to complete the questionnaires each time.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn about the quality of life, experiences with treatment, and healthcare costs of patients who are receiving long-term treatment for venous thromboembolism (VTE) that is related to cancer.

This is an investigational study. Up to 260 participants will be enrolled in this multicenter study. Up to 170 will take part in MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete 2 questionnaires either at an already-scheduled clinic visit or over the phone at the time you join this study and then about 30 days, 3 months, 6 months, and 12 months after that. These questionnaires will be about your quality of life and experiences with treatment for VTE. It should take less than 10 minutes to complete the questionnaires each time.

Information from your medical record may also be collected at these time points.

Your participation will be over after the last questionnaires are completed at about 12 months after you enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years) female or male subjects.
2. Confirmed symptomatic proximal or distal lower extremity deep venous thrombosis with or without pulmonary embolism or other venous thromboses. For a symptomatic lower extremity deep venous thrombosis confirmed by compression ultrasonography, venography, or specific computerized tomography (CT) venography, or a thrombus detected in the iliac veins on an abdominal or pelvic CT. For symptomatic pulmonary embolism confirmed by computerized tomographic pulmonary angiography, ventilation perfusion scan, or catheter pulmonary angiography.
3. Cancer (other than basal-cell or squamous-cell carcinoma of the skin), either active or diagnosed within 2 years prior to VTE. The diagnosis of cancer must be objectively documented by histopathologic diagnosis.
4. Intention for long-term treatment (at least 3 months) with anticoagulation.
5. Participants will be enrolled in the study within the first 5 days from initiation of anticoagulation.
6. Able to provide informed consent and complete study survey tools
7. Able to read and speak English.

Exclusion Criteria:

1. Indication for anticoagulation other than cancer-related VTE.
2. An Eastern Cooperative Oncology Group (ECOG) Performance Status of 4 at the time of study enrollment.
3. Life expectancy < 3 months.
4. Isolated pulmonary embolism, or isolated upper extremity deep venous thrombosis, or isolated splanchnic venous thrombosis, or isolated cerebral venous thrombosis confirmed by compression ultrasonography, venography, or CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants treated for cancer-related VTE at UT MD Anderson Cancer Center and other institutions.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Adherence to Anticoagulation | Baseline up to 6 months
  Adherence categorized as "adequate" versus "non-adequate" based on the Morisky scale.

SECONDARY OUTCOMES:
HRQL Variables in Patients for Cancer-Related VTE Treated with Anticoagulation | Baseline, 3 months, and 6 months
  The HRQL variables measured using a deep venous thrombosis quality of life questionnaire: DVTQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Cristhiam M. Rojas Hernandez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Fundacion Valle del Lili, Cali, Colombia
- Spain (2):
  - Hospital Clinic, Barcelona, Carrer de Villarroel, 170
  - Hospital German Trias i Pujol, Barcelona

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org